CLINICAL TRIAL: NCT00213044
Title: A Randomized, Controlled, Double-Blind, Cross-Over Trial of Safety, Effect on Genital Tract HIV Shedding, and Acceptability of Vaginal Use of Carraguard by HIV-Infected Women
Brief Title: A Randomized, Controlled, Cross-Over Trial of Safety of Vaginal Use of Carraguard by HIV-Infected Women
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Population Council (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); National Center for HIV STD and TB Prevention (Unknown); National Center for Infectious Diseases (Other Government); Ministry of Health, Thailand (Other Government); Chiang Rai Public Health Office (Other Government); Chiang Rai District Health Office (Other Government); Chiang Rai Municipal Health Office (Other Government); Chiang Rai Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: Population Council #316
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2017-08-15 (Actual); Status verified 2017-08

CONDITIONS: HIV Infections
Keywords: Microbicides; HIV prevention; HIV-positive women; safety; carrageenan; HIV
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Drug: Carraguard (PC-515)

SUMMARY:
Randomized, controlled, double-blinded, cross-over trial of 60 HIV-infected women recruited from general medical clinics, family planning clinics, groups/organizations working with persons living with AIDS to assess product safety, effect on genital tract HIV shedding, and product acceptability with vaginal use of Carraguard gel among HIV-infected women. Women had to be abstinent or in a seroconcordant relationship with only one partner for the study period.

DETAILED DESCRIPTION:
Carraguard™ (PC-515), the Population Council's lead candidate microbicide, was tested in a randomized, controlled trial in Chiang Rai, northern Thailand. Safety of daily product use determined by symptoms of irritation, effect on vaginal flora, vaginal epithelial disruption as determined by naked eye inspection (Day 7 and Day 14 of each arm) and colposcopic inspection on (Day 7), and other adverse effects, which may include UTI or other unforeseen problems (Day 7 and Day 14).

Genital tract HIV will be measured using samples collected by CVL (Day 7 and Day 14 of each arm) and vaginal swab (Day 7 and Day 14).

Product acceptability will be assessed through an interview-administered questionnaire once each study arm at the first follow-up visit (Day 7 of each arm), after using the product daily for 7 days.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50 years
* Plan to stay in the Chiang Rai area for at least four months
* HIV-infected, confirmed by Elisa and Western Blot tests
* Either has 1) no current sex partner and is planning to be abstinent for the study duration, or 2) has only one, HIV-infected sexual partner1 who is 18 years or older and is willing to give informed consent for confirmatory HIV testing and for the participant=s enrollment in the study. Women who have a steady partner/husband who she will not see during the study period or with whom she is not sexually active will not be required to bring their partner to the clinic for HIV testing and informed consent.
* Willing and able to give informed consent
* Willing and able to comply with the study protocol, including being tested for HIV and undergoing repeated pelvic and colposcopic examinations
* Willing to have male partner asked for informed consent because he will be exposed to study product
* Regular menstrual cycles (defined as occurring every 3-5 weeks, lasting 3-5 days) for the prior 3 months; if have amenorrhea or if using depo-provera, participant must have no reported history of vaginal bleeding for the previous 3 months
* CD4 count < 5002
* Not currently taking antiretroviral medications3
* Documented Class I or Class II ("atypical cells seen, usually caused by inflammation") pap smear at screening for study participation
* In good health as determined by medical history, physical examination and results of any laboratory screening test, and the discretion of the clinical staff
* Able to achieve a score of 80% or better on true-false test of key study concepts. If women score less than 80% the first time they take the test, they may repeat the test at least one day later

Exclusion Criteria:

* CD4 count <50
* Pregnancy or desire to become pregnant in the next 3-4 months
* Delivery, miscarriage, or abortion within six weeks prior to study enrollment
* History of surgery on external genitalia, vagina or cervix in the month prior to study enrollment
* Existence of a clinically detectable genital abnormality, specifically warts or a congenital abnormality
* History of nonmenstrual vaginal bleeding with intercourse in past one month
* Current use of tampons, diaphragms, sponges, douching, or other intravaginal products. Women who are willing to abstain from using these products during the study will be included in the study.
* Concurrent participation in another trial of a vaginal product
* History of sensitivity or allergy to latex products (including gloves)
* Presence of epithelial disruption of the labia or genital mucosa visible to the naked eye at enrollment1
* Positive test for gonorrhea, chlamydial infection, trichomoniasis, or evidence of untreated syphilis (see section 5.19). Participants with positive tests must be treated and have a negative test of cure to be eligible for enrollment.1
* Positive tests for candidiasis or bacterial vaginosis (BV) and symptoms of vaginitis. Women may be enrolled after treatment if they are asymptomatic or have negative tests. Asymptomatic participants with positive tests for candidiasis or BV may be enrolled.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60
Dates: Start 2003-03 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Safety: irritation, effect on vaginal flora, vaginal epithelial disruption determined by visual inspection (Day 7, 14) and colposcopic inspection(Day 7); other adverse effects, which may include UTI or other unforeseen problems (Day 7, 14).
Genital tract HIV: measured using samples collected by CVL (Day 7, 14) and vaginal swab (Day 7, 14).
Acceptability: interview-administered questionnaire (Day 7).

CONTACTS AND LOCATIONS:
Overall Officials: Janneke van de Wijgert, PhD, Principal Investigator — Population Council; Catherine McClean, Principal Investigator — Centers for Disease Control and Prevention
Locations (1):
- Chiang Rai Health Club, Chiang Rai, Thailand

REFERENCES:
- [Derived] Whitehead SJ, McLean C, Chaikummao S, Braunstein S, Utaivoravit W, van de Wijgert JH, Mock PA, Siraprapasiri T, Friedland BA, Kilmarx PH, Markowitz LE. Acceptability of Carraguard vaginal microbicide gel among HIV-infected women in Chiang Rai, Thailand. PLoS One. 2011;6(9):e14831. doi: 10.1371/journal.pone.0014831. Epub 2011 Sep 7. PMID 21915249
- [Derived] McLean CA, van de Wijgert JH, Jones HE, Karon JM, McNicoll JM, Whitehead SJ, Braunstein S, Achalapong J, Chaikummao S, Tappero JW, Markowitz LE, Kilmarx PH. HIV genital shedding and safety of Carraguard use by HIV-infected women: a crossover trial in Thailand. AIDS. 2010 Mar 13;24(5):717-22. doi: 10.1097/QAD.0b013e328333bf89. PMID 20098295